CLINICAL TRIAL: NCT01235585
Title: Phase III, Multi-center, Randomized, 12-week, Double-blind, Parallel-group, Placebo-controlled Study to Evaluate the Efficacy and Safety of RO4917838 in Patients With Sub-optimally Controlled Symptoms of Schizophrenia Treated With Antipsychotics Followed by a 40-week Double-blind, Parallel-group, Placebo-controlled Treatment Period.
Brief Title: A Study of RO4917838 (Bitopertin) in Patients With Sub-optimally Controlled Symptoms of Schizophrenia (WN25306)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WN25306; 2010-020616-11
Record Dates: First submitted 2010-10-22; First posted 2010-11-05 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — (4-(3-fluoro-5-trifluoromethylpyridin-2-yl)piperazin-1-yl)(5-methanesulfonyl-2-(2,2,2-trifluoro-1-methylethoxy)phenyl)methanone

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Bitopertin oral dose level 1 (Experimental)
  Interventions: Drug: bitopertin [RO4917838]
- Bitopertin oral dose level 2 (Experimental)
  Interventions: Drug: bitopertin [RO4917838]
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Oral doses, once a day for 52 weeks
  Arms: Placebo
Drug: bitopertin [RO4917838] — Oral dose level 1, once a day for 52 weeks
  Arms: Bitopertin oral dose level 1
Drug: bitopertin [RO4917838] — Oral dose level 2, once a day for 52 weeks
  Arms: Bitopertin oral dose level 2

SUMMARY:
This randomized, multi-center, double-blind, parallel-group, placebo-controlled study will evaluate the efficacy and safety of RO4917838 (bitopertin) in patients with sub-optimally controlled symptoms of schizophrenia. Patients, on stable treatment with antipsychotics, will be randomized to receive daily oral doses of RO4917838 or matching placebo for 52 weeks, followed by an optional treatment extension for up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/= 18 years of age
* Diagnosis of schizophrenia
* Clinical stability for 16 weeks (4 months) prior to randomization
* Antipsychotic treatment stability for the past 12 weeks prior to randomization
* With the exception of clozapine, patients are on any of the available marketed atypical or typical antipsychotic (treatment with a maximum of two antipsychotics)

Exclusion Criteria:

* Has treatment resistant schizophrenia as judged by the treating physician OR have failed two trials
* Evidence that patient has clinically significant uncontrolled or unstable medical disorder (e.g. cardiovascular, renal hepatic, gastrointestinal, hematologic, immunological, neurological, endocrine, metabolic or pulmonary disease)
* Patient has a body mass index (BMI) of <17 or >40 kg/m2, respectively)
* Diagnosis of mental retardation or severe organic brain syndromes
* In the investigator's judgment, a significant risk of suicide or violent behavior

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 597 (Actual)
Dates: Start 2010-12; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Positive symptoms factor score assessed by Positive and Negative Syndrome Scale (PANSS) | Change from baseline to Week 12
Safety (incidence of adverse events) | Week 12

SECONDARY OUTCOMES:
Symptom domains of schizophrenia using Positive and Negative Syndrome Scale (PANSS) | Change from baseline to Week 12
Disease improvement on Clinical Global Impression - Improvement (CGI-I) symptoms scale | Change from baseline to Week 12
Disease severity on Clinical Global Impression - Severity (CGI-S) symptoms scale | Change from baseline to Week 12
Safety (incidence of adverse events) | 60 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (94):
- United States (22):
  - Carson, California
  - Garden Grove, California
  - Long Beach, California
  - Oceanside, California
  - San Diego, California
  - Hartford, Connecticut
  - Norwalk, Connecticut
  - North Miami, Florida
  - Atlanta, Georgia
  - Chicago, Illinois
  - Hoffman Estates, Illinois
  - Joliet, Illinois
  - Lake Charles, Louisiana
  - St Louis, Missouri
  - Omahac, Nebraska
  - Cedarhurst, New York
  - Jamaica, New York
  - Rochester, New York
  - Allentown, Pennsylvania
  - Norristown, Pennsylvania
  - Philadelphia, Pennsylvania
  - Bothell, Washington
- Brazil (9):
  - Salvador, Estado de Bahia
  - Goiânia, Goiás
  - Belo Horizonte, Minas Gerais
  - Curitiba, Paraná
  - Rio de Janeiro, Rio de Janeiro
  - Pelotas, Rio Grande do Sul
  - Porto Alegre, Rio Grande do Sul
  - Itapira, São Paulo
  - São Paulo, São Paulo
- Canada (8):
  - Calgary, Alberta
  - Medicine Hat, Alberta
  - Vancouver, British Columbia
  - Halifax, Nova Scotia
  - Burlington, Ontario
  - Hamilton, Ontario
  - Mississauga, Ontario
  - Montreal, Quebec
- Chile (2):
  - Santiago
  - Valdivia
- Germany (7):
  - Berlin
  - Bochum
  - Cologne
  - Freiburg im Breisgau
  - Hamburg
  - München
  - Nuremberg
- Latvia (3):
  - Daugovpils
  - Jelgava
  - Liepāja
- Lithuania (3):
  - Kaunas
  - Šilutė
  - Vilnius
- Netherlands (2):
  - Assen
  - Groningen
- Poland (7):
  - Choroszcz
  - Kielce
  - Lublin
  - Piekary Śląskie
  - Skorzewo
  - Tuszyn
  - Warsaw
- Slovakia (5):
  - Bojnice
  - Bratislava
  - Rimavská Sobota
  - Svidník
  - Trnava
- Spain (5):
  - Barcelona, Barcelona
  - Madrid, Madrid
  - Oviedo, Principality of Asturias
  - Salamanca, Salamanca
  - Zamora, Zamora
- Taiwan (6):
  - Hualian Town
  - Kaohsiung City
  - Taichung
  - Tainan
  - Tainan County
  - Taipei
- Turkey (Türkiye) (7):
  - Ankara
  - Diyarbakır
  - Gaziantep
  - Istanbul
  - Kocaeli
  - Manisa
  - Mersin
- Ukraine (8):
  - Dnipropetrovsk
  - Donetsk
  - Glevakha Kyviv Region
  - Kharkiv
  - Kyiv
  - Lviv
  - Odesa
  - Vinnytsia

REFERENCES:
- [Derived] Bugarski-Kirola D, Iwata N, Sameljak S, Reid C, Blaettler T, Millar L, Marques TR, Garibaldi G, Kapur S. Efficacy and safety of adjunctive bitopertin versus placebo in patients with suboptimally controlled symptoms of schizophrenia treated with antipsychotics: results from three phase 3, randomised, double-blind, parallel-group, placebo-controlled, multicentre studies in the SearchLyte clinical trial programme. Lancet Psychiatry. 2016 Dec;3(12):1115-1128. doi: 10.1016/S2215-0366(16)30344-3. Epub 2016 Nov 2. PMID 27816567